CLINICAL TRIAL: NCT04210960
Title: Correlation of Serum Lactate and Activity of Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Esmael, Assistant Prof of Neurology, Mansoura University Hospital
Other Study IDs: Mansoura University H 10
Record Dates: First submitted 2019-12-22; First posted 2019-12-26 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis, serum lactate and MRS
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients group: 50 multiple sclerosis patients
  Interventions: Radiation: Magentic resonanace imaging; Radiation: Magentic resonanace spectroscopy
- Control group: 30 normal healthy control
  Interventions: Radiation: Magentic resonanace imaging; Radiation: Magentic resonanace spectroscopy

INTERVENTIONS:
Radiation: Magentic resonanace imaging — The brain MR imaging examinations were done by using a 3 tesla scanner (Acheiva; Philips Medical Systems, Best, Netherlands). All patients were examined in the supine position using head coil. Routine images (T2, T1, FLAIR) and double inversion recovery sequence (DIR) were done to all patients: repetition time (TR) _ 9583 sec, echo time (TE) _ 25 sec, inversion time (TI) _ 3400 sec, IR delay _ 325 sec, echo train length (ETL) _ 17, 50 contiguous axial slices, thickness _ 3 mm, matrix size 240× 142 mm2, field of view (FOV) 230× 184 mm2.
Radiation: Magentic resonanace spectroscopy — Magnetic Resonance (MR) spectroscopy is a noninvasive diagnostic test for measuring biochemical changes in the brain.While magnetic resonance imaging (MRI) identifies the anatomical location of a lesion, MR spectroscopy compares the chemical composition of normal brain tissue with abnormal brain tissue. This test can also be used to detect tissue changes in stroke and epilepsy.

SUMMARY:
Correlation of serum lactate and activity of multiple sclerosis and its correlation to different type of MS

DETAILED DESCRIPTION:
Correlation of serum lactate and activity of multiple sclerosis and its correlation to different type of MS and magentic resonanace imaging , magentic resonanace spectroscopy

ELIGIBILITY:
Inclusion Criteria:

-Patients with multiple sclerosis (RRMS,PPMS and SPMS)

Exclusion Criteria:

-Patients with any other medical conditions that may affect the serum lactate level

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 80 Egyptian subjects (50 multiple sclerosis patients (patients group = group I) and 30 normal healthy control (control group = group II)
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-12-23 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Biochemical testing | 2 days
  Plasma lactate was assayed according to Trinder method14 . All assays were carried out with Bechman Coulter AU480 autoanalyzer (USA).

CONTACTS AND LOCATIONS:
Overall Officials: Esmael M Ahmed, MD, Principal Investigator — Assistant Prof of Neurology
Locations (1):
- Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Esmael A, Talaat M, Egila H, Eltoukhy K. Mitochondrial dysfunction and serum lactate as a biomarker for the progression and disability in MS and its correlation with the radiological findings. Neurol Res. 2021 Jul;43(7):582-590. doi: 10.1080/01616412.2021.1893567. Epub 2021 Mar 4. PMID 33657991